CLINICAL TRIAL: NCT06764004
Title: The Effect of Human Umbilical Cord Mesenchymal Stem Cells and Exosomes on the Healing of Postoperative Pain and Periapical Lesions in the Treatment of Apical Periodontitis: Randomized Controlled Clinical Study
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ipek Eraslan Akyuz, Dentist, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025
Record Dates: First submitted 2024-12-22; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Apical Periodontitis
Keywords: Regenerative endodontics, rejeneration, stem cell
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Stem cell group (Experimental): Human umbilical cord stem cells will be used.
  Interventions: Genetic: Stem Cell Product
- Exosome group (Experimental): Exosomes obtained from umbilical cord stem cells will be used.
  Interventions: Genetic: Stem Cell Product
- Bleeding group (Experimental): A clot will be formed by bleeding in the periapical region of the root canals.
  Interventions: Biological: Bleeding and clots

INTERVENTIONS:
Genetic: Stem Cell Product — Human umbilical cord stem cells and exosomes will be used.
  Arms: Exosome group; Stem cell group
Biological: Bleeding and clots — Exosomes obtained from human umbilical cord stem cells will be used
  Arms: Bleeding group

SUMMARY:
The main purpose of this study is to evaluate the effect of Mesenchymal Stem Cells (MSCs) isolated from the umbilical cord and exosomes derived from these cells on the success of the treatment in the regenerative endodontic treatment of necrotic open apex molar teeth.

Regenerative endodontic treatment aims to disinfect root canals and revascularize pulp tissue. Our goals in this study are; obtaining umbilical cord-derived MSCs, obtaining exosomes derived from umbilical cord MSCs, selecting patients with molar teeth with necrotic open apex and periapical lesion, initiation of regenerative endodontic treatment and disinfection of root canals, induction of bleeding in the periapical region and formation of a blood clot in the root canal in the 1st patient group, in the 2nd patient group, umbilical cord-derived MSCs were placed in the root canals without bleeding in the periapical region, in the 3rd patient group, placement of exosomes from umbilical cord-derived MSCs into the root canals without causing bleeding in the periapical region, it is the follow-up of patients at regular intervals for up to 1 year after treatment is completed.

DETAILED DESCRIPTION:
Endodontic treatment of immature, permanent teeth is one of the most challenging situations encountered in endodontics. The dentin walls of the roots of these teeth are thin and fragile, making it difficult to properly clean, prepare and fill. In immature permanent teeth, pulp necrosis causes root development to stop and the apex to remain open. Etiology of pulp necrosis; It may be due to caries, trauma or the presence of dental anomalies (dens invaginatus and dens evaginatus). Today, there is a paradigm shift in the treatment of such cases from traditional apexification procedures to regenerative endodontic procedures. The aim of both treatments is; The aim is to cure apical pathology, eliminate symptoms, stimulate root development by closing the apical opening, and restore the functional adequacy of the pulp tissue. Regenerative endodontic therapy involves procedures designed to repair or replace damaged tooth structures or regenerate part of the pulp-dentin complex. Many studies have shown that this treatment can achieve positive results, leading to resolution of the patient's initial signs and symptoms, complete healing of periapical tissues, thickening of the root canal wall, and continued root maturation with apical closure. The success of regenerative endodontic treatments depends on the presence of three critical components: a- Mesenchymal stem cells that form the source of odontoblast-like cells, b- Growth factors required for the stimulation, differentiation and proliferation of mesenchymal stem cells (MSCs), and c- A suitable environment for the continuation of root development. A physical scaffolding that provides an environment. With this treatment, undifferentiated mesenchymal cells replace the dentin and pulp tissue and the development of the roots continues. In addition, a positive response to viability tests can be achieved in teeth by causing bleeding in the periapical tissues. In a study conducted by Lovelace et al., they revealed that a significant amount of stem cells could be stimulated by induction of bleeding in the periapical region after disinfection of root canals. Many case reports have demonstrated that regenerative endodontic procedures using blood clots show successful results. Nowadays, various researchers aim to create more current regenerative therapy procedures using new biomaterials for the regeneration of tissues. Many approaches can be combined using different stem cells, scaffolds and growth factors to regenerate or repair teeth and supporting tissues.

MSCs are multipotent cells with low immunogenic potential that can be isolated from tissues such as bone marrow, adipose tissue and umbilical cord. Bone marrow-derived MSCs have generally been used in many experimental and clinical studies, but obtaining these cells has some disadvantages such as requiring invasive procedures and a reduced proliferation and differentiation potential associated with donor age and concomitant diseases. In contrast, umbilical cord-derived MSCs are easily obtainable and have higher differentiation potential. The therapeutic potential of umbilical cord-derived stem cells to treat a wide variety of disorders has led to their increased use in the treatment of many diseases, including regenerative therapy and modulation of refractory autoimmune diseases. In a study by Sun et al. evaluating the effectiveness of human umbilical cord MSC infusion in children with autism spectrum disorder, improvements in autism symptoms were reported. In the study by Brizuela et al., in which the effectiveness of using allogeneic umbilical cord stem cells in the regenerative treatment of teeth with periapical lesions was evaluated, it was reported that there was a reduction in the size of the apical lesion and a positive response was obtained from the teeth in sensitivity tests.

Exosomes are extracellular vesicles with different sizes ranging from 30-200 nm in diameter. Exosomes have been found to be secreted by many cell types, including immune system cells, neuronal, epithelial, endothelial, embryonic cells, and MSCs. Exosomes may contain various types of vesicles, including microvesicles and apoptotic bodies. Similarly, recent studies on the effectiveness of MSC-derived exosomes have found that they may have advantageous effects in a variety of contexts, including respiratory, cartilage, kidney, heart and liver diseases, bone repair and cancer. In a review study by Hammouda et al., it was reported that the use of stem cell-derived exosomes in regenerative therapies could be a promising regenerative tool for dentin-pulp complex regeneration.

Considering the literature information compiled above, the aim of this study is to evaluate the effect of human umbilical cord MSCs and exosomes on the healing of postoperative pain and periapical lesions through clinical and radiographic examinations in the regenerative endodontic treatment of necrotic open apex molar teeth.

ELIGIBILITY:
Inclusion Criteria:

1. Molar teeth with open apex
2. Teeth with apical periodontitis
3. Teeth for which prosthetic restoration is not planned
4. Patients between the ages of 9-15 without any significant health problems
5. Patients who are not accompanied by periodontal problems and whose oral hygiene is in good condition

Exclusion Criteria:

1. Individuals with systemic diseases and allergic reactions
2. Severely damaged teeth
3. Previous root canal treatment has been performed on the tooth.
4. Use of antibiotics, anti-inflammatory, and painkillers in the last two weeks
5. Teeth with cracks and broken lines

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of patients' postoperative pain with a questionnaire | 1-4 months
  It indicates the achievement of outcome measures upon completion of the treatment administered to patients. Pain assessment will be made with the visual analog scale (VAS). A score between 0 and 100 will be given for pain evaluation. '0' indicates no pain, '100' indicates severe pain.

SECONDARY OUTCOMES:
Follow-up of patients with questionnaire their pain and symptoms at regular intervals for up to 1 year | 1-12 mouths
  Completion of the follow-up period of patients after regenerative endodontic treatment indicates that the secondary outcome measures have been achieved. Pain assessment will be made with the visual analog scale (VAS). A score between 0 and 100 will be given for pain evaluation. '0' indicates no pain, '100' indicates severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Melikgazi, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No